CLINICAL TRIAL: NCT01964183
Title: Post-Marketing Study of Mirabegron - A Pharmacokinetic Study to Assess Drug-Drug Interaction Between Mirabegron and Tolterodine -
Brief Title: Post-marketing Study to Evaluate the Effect of Mirabegron on the Plasma Concentration of Tolterodine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 178-CL-111
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2013-10-17 (Estimated); Status verified 2013-10

CONDITIONS: Pharmacokinetics of Mirabegron and Tolterodine; Healthy
Keywords: Open-label design; Pharmacokinetics; Drug-Drug Interaction; Mirabegron
MeSH Terms: interventions — Tolterodine Tartrate; mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- treatment group (Experimental)
  Interventions: Drug: tolterodine; Drug: mirabegron

INTERVENTIONS:
Drug: tolterodine — Oral
  Other Names: Detrusitol® Capsules
Drug: mirabegron — Oral
  Other Names: YM178; Betanis® tablets

SUMMARY:
To assess the effect of multiple doses of mirabegron to postmenopausal adult female subjects on the pharmacokinetics (PK) of tolterodine and its metabolites.

In addition, the safety of these products will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of two years after menopause
* Body weight (at screening) ≥ 40.0 kg and < 70.0 kg
* Body mass index (BMI) (at screening) ≥ 17.6 kg/m2 and < 26.4 kg/m2
* Healthy, as judged by the investigator/sub-investigator based on medical history and the results of physical examination (subjective symptoms and objective findings) and all tests obtained at screening and during the period from hospital admission (at single dosing phase) to immediately before study medication.

Exclusion Criteria:

* Received or scheduled to receive any investigational drugs in other clinical trials, post-marketing studies, or clinical studies within 120 days before the screening or during the period from the screening to hospitalization (Day -2).
* Donated or scheduled to donate 400 mL of whole blood within 90 days before the screening or during the period from the screening to hospitalization (Day -2), 200 mL of whole blood within 30 days before the screening or during the period from the screening to hospitalization (Day -2), or blood components within 14 days before the screening or during the period from the screening to hospitalization (Day -2).
* Any deviation of the laboratory tests at screening or hospitalization (Day -2).
* A deviation from the normal range of blood pressure, pulse rae, or body temperature at screening or hospitalization (Day -2) Supine blood pressure: Systolic blood pressure: ≥90 mmHg, ≤140 mmHg, Diastolic blood pressure: ≥40 mmHg, ≤90 mmHg Supine pulse rate; ≥40 bpm, ≤99 bpm Axillary body temperature; ≥35.0°C, ≤37.0°C
* History of drug allergies
* Upper gastrointestinal disease (e.g., nausea, vomiting, and stomachache) within 7 days before hospitalization (Day -2)
* Concurrent or previous hepatic disease (e.g., viral hepatitis, drug-induced liver injury, and hepatic impairment)
* Concurrent or previous heart disease (e.g., congestive heart failure, angina pectoris, and arrhythmia requiring treatment)
* Concurrent or previous GI disease (e.g., ileus paralytic, gastric atony, intestinal atony, colitis ulcerative, peptic ulcer and gastroesophageal reflux esophagitis; except for a history of appendicitis).
* Concurrent or previous renal disease (e.g., acute renal failure, glomerulonephritis, and interstitial nephritis)
* Concurrent or previous endocrine disease (e.g., hyperthyroidism and blood growth hormone abnormal)
* Concurrent or previous cerebrovascular disorder (e.g., cerebral infarction)
* Previous use of mirabegron or tolterodine
* Excessive smoking or drinking habit

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of unchanged mirabegron | Day 14
Plasma concentration of unchanged tolterodine | Day 7, Day 14

SECONDARY OUTCOMES:
Plasma concentration of tolterodine metabolites (5-hydroxymethyl tolterodine; 5-HMT) | Day 7, Day 14
Safety assessed by the incidence of adverse events, vital signs, clinical labo-tests, and 12-lead ECG | Day -2, Day 8, Day 15, Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Chair — Astellas Pharma Inc
Locations (1):
- Kanto, Japan